CLINICAL TRIAL: NCT03718156
Title: The Prevention Program for Alzheimer's Related Delirium (PREPARED) Cluster Randomized Trial
Brief Title: The Prevention Program for Alzheimer's Related Delirium (PREPARED) Trial
Acronym: PREPARED
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented us from continuing this study which involves active participation from long-term care front-line staff. More funding is being sought to continue our trial
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Machelle Wilchesky, Assistant Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PT 71435
Record Dates: First submitted 2018-08-20; First posted 2018-10-24 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Delirium; Dementia
Keywords: delirium; dementia; long-term care; cluster randomized trial; nursing; geriatrics
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Intervention Model Description: The PREPARED Trial is a 4-year cluster randomized intervention study. A cluster design was adopted in order to prevent contamination across the intervention and control arms by nursing staff who may provide replacement hours of employment at different units/floors within their long-term care facilities (LTCFs). Participating LTCFs (clusters) will be assigned to either the PREPARED Trial intervention or the control (usual care) arm of the study using a covariate constrained randomization procedure. In addition, given the need to assess each resident weekly for a follow-up period of 18 weeks and logistical limitations (large geographical coverage, 40-50 LTCFs included, and limited work force), the investigators will employ a sequential approach whereby sets of clusters (LTCFs) will be randomized into the two study arms in consecutive 'waves' of follow-up lasting 18 weeks each. It is estimated that 4 waves of trial follow-up, comprised of 10-12 clusters each, will be completed.
Masking Description: Long-term care facilities (LTCFs) cannot be blinded, as trial arm allocation will be obvious (those in the intervention group will undergo delirium prevention protocol training before their respective follow-up periods, and those in the control group will not). Similarly, research assistants (RAs) tasked with conducting resident assessments cannot be blinded to group allocation, as they will be constantly exposed to the everyday workings of participating LTCFs. However, RAs will be blinded to resident cognitive scores. All researchers analyzing the data will be blinded to group allocation, as LTCF names will be anonymized and randomization statuses will be concealed prior to data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREPARED Trial Intervention (Experimental): Participating nursing staff will be trained to apply the PREPARED Trial interventions, and will apply this knowledge to modify the therapeutic nursing plans of residents under their care who are enrolled in the study, accordingly.
  Interventions: Other: PREPARED Trial Intervention
- Care as Usual (No Intervention): Participating nursing staff will only be provided with general information about delirium, but will not be trained or instructed to modify the therapeutic nursing plans that are in place for residents enrolled in the study. However, at the end of the follow-up period, nursing staff in the control arm will be provided with the PREPARED Trial intervention training program (including bedside coaching), which they can then use after the study has ended at their facility.

INTERVENTIONS:
Other: PREPARED Trial Intervention — Nursing staff members will be trained to adjust the therapeutic nursing plans (TNP) for residents enrolled in the study, as follows: 1) by providing optimal stimulation (surveying the use of eyeglasses and hearing aids, the room lighting and space organization; orienting the resident to time and space; and stimulating the resident using familiar objects, photos, and life histories); and 2) by assessing the presence of 4 modifiable delirium risk factors (antipsychotic use, sensory impairment, restraint use, and dehydration) and taking specific actions once a given risk factor is identified. For instance, if physical restraints are used, the TNP will require that they are to be removed during care when a caregiver is present (nail care, feeding, and wound care).
  Arms: PREPARED Trial Intervention

SUMMARY:
By the year 2038, over a million Canadians are expected to have Alzheimer's disease, a type of dementia. Dementia increases the risk of nursing home placement among the elderly more than fivefold. Given the exceptionally vulnerable nature of this patient population, there is a pressing need to ensure that the clinical care they receive is evidence-based, tailored specifically for them, and meeting the high standards of quality that would be expected in any other health-care setting. Delirium is a sudden and severe change in brain function that can cause a person to appear confused or disoriented, have memory loss, and have difficulties maintaining focus. It is an urgent care issue facing elderly patients residing in nursing homes, or long-term care (LTC) facilities. Delirium is a significant cause of illness and mortality, affecting between 10%-89% of LTC patients, but little research has focused on delirium prevention in the LTC setting. This study will assess the effectiveness of a LTC multicomponent delirium prevention program (PREPARED Trial intervention). The PREPARED Trial intervention is an intervention provided to nursing staff working in LTC facilities that consists of four components: a decision tree, an instruction manual, a training package, and a toolkit. The feasibility and acceptability of the PREPARED Trial intervention has already been successfully demonstrated; however, a thorough and well-designed large scale study is needed in order to confirm its ability to reduce delirium among LTC residents. In this study, approximately 40-50 LTC facilities will be randomized to either receive the PREPARED Trial intervention or to receive usual care. At the end of the 4-year study period, the investigators will be able to demonstrate the degree to which the PREPARED Trial intervention reduces: 1) the number of new cases of delirium; 2) delirium severity; and 3) the duration of delirium episodes. This study will provide the blueprint of a program that can be transferable to LTC facilities across Canada.

DETAILED DESCRIPTION:
Overall Goal: To reduce the incidence, severity, duration, and frequency of delirium episodes in cognitively impaired long-term care (LTC) residents at high risk for delirium.

Background: Delirium is a significant cause of morbidity and mortality among older people admitted to both acute and LTC settings. Prevention, founded on a thorough understanding of associated risk factors, is the best approach for dealing with delirium. Several successful multicomponent interventions have been developed to reduce delirium incidence in the acute care setting (30%-73% reduction) by intervening on identified modifiable risk factors. Little work, however, has focused on using this approach to reduce delirium incidence in LTC. As such, co-investigators within the study team employed an integrated knowledge translation strategy to develop a LTC multicomponent delirium prevention program (PREPARED Trial intervention). The feasibility and acceptability of this program has been demonstrated using a participatory approach in two Quebec LTC facilities (LTCFs), and the program has received recognition by the scientific community. Given its large expected impact and high knowledge translation potential, a thorough and well-designed large-scale evaluation is urgently needed in order to demonstrate the effectiveness of the multicomponent delirium prevention program in preventing delirium among high-risk LTC residents.

Primary Objective: To assess efficacy of the PREPARED Trial intervention in reducing delirium incidence, and delirium episode severity, duration, and frequency among cognitively impaired, high-risk LTC residents.

Secondary Objectives: To compare the effect of the PREPARED Trial intervention to that of usual care on the incidence of falls among cognitively impaired LTC residents, to estimate the association between medication use and delirium incidence in LTCFs, to estimate if there is an effect modification by motor subtype of delirium or by dementia subtype, and to measure the prevalence of delirium in participating institutions.

Tertiary Objectives: To compare the effect of the PREPARED Trial intervention on other health outcomes, including: changes in functional autonomy or social engagement, the number of transfers to acute care, consultations with healthcare providers, and mortality rates.

Methods: This 4-year cluster randomized study will involve nursing staff and residents in 40-50 public and semi-private LTC facilities in Quebec, Canada. Institutions within all 5 of the Montreal island Integrated University Health and Social Services networks (CIUSSS) and one private provincial network are currently participating. Approximately 900 LTC residents will be enrolled in the study and followed for 18 weeks only if they are at high risk of delirium and are delirium-free at baseline. The PREPARED Trial intervention is a program consisting of four components: a decision tree, an instruction manual, a training package and a toolkit. Primary study outcomes such as delirium incidence (measured by the Confusion Assessment Method), delirium severity (measured by the Delirium Index), and level of adherence to the PREPARED Trial protocol will be assessed weekly. Functional autonomy levels will be assessed at the beginning and end of follow-up, while information pertaining to modifiable delirium risk factors, medical consultations, and institutional transfers will be collected for the duration of the follow-up period. For primary analysis, hazard ratios will be modeled using Cox regression to compare the effect of the PREPARED Trial intervention to that of usual care on the time to first delirium episode. Clustering effects will be taken into account using frailty models, an extension of Cox regression for the addition of random effects.

Expected Outcomes and Significance: This large-scale intervention study will contribute significantly to the development of evidence-based clinical guidelines for delirium prevention in this frail elderly population, as it will be the first to evaluate the efficacy of a multicomponent delirium prevention program translated into LTC clinical practice on a large scale. In addition to reducing delirium in this frail population, deliverables include validation of this prevention program, as well as the transferring of its components (including bilingual video training modules for LTC staff) to relevant knowledge users across Canada.

ELIGIBILITY:
Inclusion Criteria:

* has dementia and/or cognitive impairment (as determined by discussions with the nursing staff and chart abstraction);
* a minimum length of stay in the LTC institution of at least two weeks prior to the start of the baseline assessments;
* at high risk of delirium, as indicated by a score of 3 or higher on a validated 5-item delirium risk screening tool;
* delirium-free at baseline, as assessed by the Confusion Assessment Method (CAM), the Delirium Index (DI) and a brief chart review over a screening period of two consecutive weeks.

Exclusion Criteria:

* unable to communicate verbally in English or French (as determined by either the nursing staff or two consecutive 0-score administrations of the composite cognitive interview at screening);
* has a history of specific psychiatric conditions (bipolar disorder, depression with signs of psychosis, and psychotic disorders) or intellectual disability;
* is receiving comfort/end-of-life care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-06-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | over the 18 week follow-up period
  Confusion Assessment Method (CAM) scores
Delirium severity | over the 18 week follow-up period
  Delirium Index scores (0-21)
Delirium episode duration | over the 18 week follow-up period
  the total number of days that a given resident experiences active episode(s) of delirium
Number of delirium episodes | over the 18 week follow-up period
  count of delirium episodes

SECONDARY OUTCOMES:
Delirium motoric subtype | over the 18 week follow-up period
  Delirium Motor Subtype Scale scores
Number of falls | over the 18 week follow-up period
  count of falls and fall-related injuries, as documented in medical charts
Time to first fall | over the 18 week follow-up period
  days to first reported fall
Change in functional autonomy | over the study period (18 weeks)
  Barthel Index (Shah version) scores
Change in cognitive functioning | over the study period (18 weeks)
  Hierarchic Dementia Scale scores
Change in level of social engagement | over the study period (18 weeks)
  Revised Index of Social Engagement in Long-Term Care Facilities scores

CONTACTS AND LOCATIONS:
Overall Officials: Machelle Wilchesky, PhD, Principal Investigator — McGill University; Philippe Voyer, Inf. PhD, Study Chair — Laval University; Nathalie Champoux, MD, MSc, Study Chair — Université de Montréal; Antonio Ciampi, PhD, Study Chair — McGill University; Ovidiu Lungu, PhD, Study Chair — Université de Montréal; Jane McCusker, MD, PhD, Study Chair — McGill University; Johanne Monette, MD, MSc, Study Chair — Lady Davis Institute for Medical Research; T.T. Minh Vu, MD, FRCPC, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (6):
- Canada (6):
  - Association des établissements privés conventionnés, Montreal
  - Integrated University Health and Social Services Centre for East Montreal, Montreal
  - Integrated University Health and Social Services Centre for North Montreal, Montreal
  - Integrated University Health and Social Services Centre for South-Central Montreal, Montreal
  - Integrated University Health and Social Services Centre for West Montreal, Montreal
  - Integrated University Health and Social Services Centre for West-Central Montreal, Montreal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elie M, Rousseau F, Cole M, Primeau F, McCusker J, Bellavance F. Prevalence and detection of delirium in elderly emergency department patients. CMAJ. 2000 Oct 17;163(8):977-81. PMID 11068569
- [Background] Fick DM, Agostini JV, Inouye SK. Delirium superimposed on dementia: a systematic review. J Am Geriatr Soc. 2002 Oct;50(10):1723-32. doi: 10.1046/j.1532-5415.2002.50468.x. PMID 12366629
- [Background] Lemiengre J, Nelis T, Joosten E, Braes T, Foreman M, Gastmans C, Milisen K. Detection of delirium by bedside nurses using the confusion assessment method. J Am Geriatr Soc. 2006 Apr;54(4):685-9. doi: 10.1111/j.1532-5415.2006.00667.x. PMID 16686883
- [Background] Voyer P, Richard S, Doucet L, Carmichael PH. Detecting delirium and subsyndromal delirium using different diagnostic criteria among demented long-term care residents. J Am Med Dir Assoc. 2009 Mar;10(3):181-8. doi: 10.1016/j.jamda.2008.09.006. Epub 2009 Jan 8. PMID 19233058
- [Background] McCusker J, Cole MG, Voyer P, Monette J, Champoux N, Ciampi A, Vu M, Belzile E. Prevalence and incidence of delirium in long-term care. Int J Geriatr Psychiatry. 2011 Nov;26(11):1152-61. doi: 10.1002/gps.2654. Epub 2011 Jan 27. PMID 21274904
- [Background] Cole MG. Persistent delirium in older hospital patients. Curr Opin Psychiatry. 2010 May;23(3):250-4. doi: 10.1097/YCO.0b013e32833861f6. PMID 20224406
- [Background] Cole MG, McCusker J. Treatment of delirium in older medical inpatients: a challenge for geriatric specialists. J Am Geriatr Soc. 2002 Dec;50(12):2101-3. doi: 10.1046/j.1532-5415.2002.50634.x. No abstract available. PMID 12473034
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Reston JT, Schoelles KM. In-facility delirium prevention programs as a patient safety strategy: a systematic review. Ann Intern Med. 2013 Mar 5;158(5 Pt 2):375-80. doi: 10.7326/0003-4819-158-5-201303051-00003. PMID 23460093
- [Background] Vidan MT, Sanchez E, Alonso M, Montero B, Ortiz J, Serra JA. An intervention integrated into daily clinical practice reduces the incidence of delirium during hospitalization in elderly patients. J Am Geriatr Soc. 2009 Nov;57(11):2029-36. doi: 10.1111/j.1532-5415.2009.02485.x. Epub 2009 Sep 15. PMID 19754498
- [Background] Hshieh TT, Yue J, Oh E, Puelle M, Dowal S, Travison T, Inouye SK. Effectiveness of multicomponent nonpharmacological delirium interventions: a meta-analysis. JAMA Intern Med. 2015 Apr;175(4):512-20. doi: 10.1001/jamainternmed.2014.7779. PMID 25643002
- [Background] Martinez F, Tobar C, Hill N. Preventing delirium: should non-pharmacological, multicomponent interventions be used? A systematic review and meta-analysis of the literature. Age Ageing. 2015 Mar;44(2):196-204. doi: 10.1093/ageing/afu173. Epub 2014 Nov 25. PMID 25424450
- [Background] Gentric A, Le Deun P, Estivin S. [Prevention of delirium in an acute geriatric care unit]. Rev Med Interne. 2007 Sep;28(9):589-93. doi: 10.1016/j.revmed.2007.04.004. Epub 2007 May 15. French. PMID 17512095
- [Background] Pisani MA, Murphy TE, Van Ness PH, Araujo KL, Inouye SK. Characteristics associated with delirium in older patients in a medical intensive care unit. Arch Intern Med. 2007 Aug 13-27;167(15):1629-34. doi: 10.1001/archinte.167.15.1629. PMID 17698685
- [Background] Voyer P, McCusker J, Cole MG, Monette J, Champoux N, Vu M, Ciampi A, Sanche S, Richard S, de Raad M. Feasibility and acceptability of a delirium prevention program for cognitively impaired long term care residents: a participatory approach. J Am Med Dir Assoc. 2014 Jan;15(1):77.e1-9. doi: 10.1016/j.jamda.2013.08.013. Epub 2013 Oct 2. PMID 24094898
- [Background] Rockwood K. Making delirium prevention acceptable in nursing homes. J Am Med Dir Assoc. 2014 Jan;15(1):6-7. doi: 10.1016/j.jamda.2013.09.002. Epub 2013 Oct 8. No abstract available. PMID 24113630
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008 May;56(5):823-30. doi: 10.1111/j.1532-5415.2008.01674.x. Epub 2008 Apr 1. PMID 18384586
- [Background] McCusker J, Cole MG, Dendukuri N, Belzile E. The delirium index, a measure of the severity of delirium: new findings on reliability, validity, and responsiveness. J Am Geriatr Soc. 2004 Oct;52(10):1744-9. doi: 10.1111/j.1532-5415.2004.52471.x. PMID 15450055
- [Background] Allison PD (1995) Survival analysis using SAS: A practical guide. Cary, NC: SAS Institute. Inc.
- [Background] Klein J. ea (2003) Survival Analysis (2nd ed.). New York: Springer.
- [Background] Therneau TM, Grambsch PM (2000) Modeling survival data: extending the Cox model: Springer Science & Business Media.
- [Derived] Wilchesky M, Ballard SA, Voyer P, McCusker J, Lungu O, Champoux N, Vu TTM, Cole MG, Monette J, Ciampi A, Belzile E, Carmichael PH, McConnell T. The PREvention Program for Alzheimer's RElated Delirium (PREPARED) cluster randomized trial: a study protocol. BMC Geriatr. 2021 Nov 16;21(1):645. doi: 10.1186/s12877-021-02558-3. PMID 34784897